CLINICAL TRIAL: NCT06595498
Title: Evaluation of an Ultrasensitive Next Generation Sequencing Method for the Detection of EGFR Gene Mutations in the Plasma of Patients With Lung Cancer
Brief Title: Next Generation Sequencing Method for the Detection of EGFR Gene Mutations in the Plasma of Patients With Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RARE study
Record Dates: First submitted 2024-08-07; First posted 2024-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-small Cell Lung Cancer (NSCLC)
Keywords: lung cancer; non-small cell lung cancer; EGFR mutation; Next Generation Sequencing; plasma
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeqSensei™ Solid Cancer IVD Kit (Sysmex) (Experimental)
  Interventions: Diagnostic Test: Plasma- SeqSensei™ Solid Cancer IVD Kit (Sysmex)
- cobas® EGFR Mutation Test v2 (Roche) (Active Comparator)
  Interventions: Diagnostic Test: cobas® EGFR Mutation Test v2 (Roche)

INTERVENTIONS:
Diagnostic Test: Plasma- SeqSensei™ Solid Cancer IVD Kit (Sysmex) — The patients' blood has already been collected in Streck tubes for circulating DNA and the plasma has been stored at -80°C as per the procedure for the routine diagnostic test cobas EGFR Mutation Test v2. No further blood sampling will be required from patients. Circulating DNA/RNA will be extracted from 2-5 ml of plasma. The extracted cfDNA will be quantified. The libraries will be prepared using the NGS Plasma-SeqSensei™ Solid Cancer IVD Kit (Sysmex) and will be evaluated at the Tapestation (Agilent) to verify their quality and quantity using D1000 Screentapes. The libraries consisting of approximately 16 samples each will then be sequenced on an Illumina NextSeq 500 sequencer using the Illumina NextSeq 500/550 Mid Output Kit v2.5 (150 Cycles). Data analysis will be performed using Plasma-SeqSensei™ IVD Software (Sysmex).
  Arms: SeqSensei™ Solid Cancer IVD Kit (Sysmex)
Diagnostic Test: cobas® EGFR Mutation Test v2 (Roche) — The patients' blood has already been collected in Streck tubes for circulating DNA and the plasma has been stored at -80°C as per the procedure for the routine diagnostic test cobas EGFR Mutation Test v2. No further blood sampling will be required from patients. Circulating DNA/RNA will be extracted from 2-5 ml of plasma. The extracted cfDNA will be quantified. The libraries will be prepared using the cobas® EGFR Mutation Test v2 (Roche) and will be evaluated at the Tapestation (Agilent) to verify their quality and quantity using D1000 Screentapes. The libraries consisting of approximately 16 samples each will then be sequenced on an Illumina NextSeq 500 sequencer using the Illumina NextSeq 500/550 Mid Output Kit v2.5 (150 Cycles).
  Arms: cobas® EGFR Mutation Test v2 (Roche)

SUMMARY:
The study aims to evaluate the Plasma-SeqSensei™ Solid Cancer IVD Kit NGS diagnostic test (Sysmex) before its introduction into routine diagnostics. This is a test for research of EGFR mutations in cfDNA that needs to be evaluated in a patient population with lung adenocarcinoma already characterized for EGFR mutations by a molecular test of reference. The proposed study does not present any risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females aged at least 18 years;
* Patients with advanced or metastatic non-small cell lung cancer at diagnosis or progression who have previously had the cobas® EGFR Mutation Test v2 (Roche) performed on a liquid biopsy with a valid result (positive or negative);
* Availability of 6 mL of plasma.

Exclusion Criteria:

* Plasma not available in sufficient quantities to perform both tests;
* Cobas test with invalid result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Through study completion, an average of 1 year
  Evaluate the capability of the NGS test Plasma-SeqSensei™ Solid Cancer IVD Kit (Sysmex) in detecting a greater number of EGFR mutations compared to the diagnostic test routine cobas® EGFR Mutation Test v2 (Roche)

SECONDARY OUTCOMES:
Secondary Outcome | Through study completion, an average of 1 year
  Check if the NGS Plasma-SeqSensei™ Solid Cancer IVD Kit (Sysmex) is comparable to conventional test (cobas® EGFR MutationTest v2 (Roche)) in the detection of the mutational status of EGFR

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy

IPD SHARING:
Plan to Share IPD: No